CLINICAL TRIAL: NCT02349477
Title: Gabapentin for Relapse Prevention: Alcohol Withdrawal Effects
Brief Title: Gabapentin for Alcohol Relapse Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00032587
Record Dates: First submitted 2015-01-15; First posted 2015-01-29 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Alcohol Use Disorder; Alcohol Withdrawal
MeSH Terms: conditions — Alcoholism | interventions — Gabapentin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin (Experimental): Gabapentin up to 1200 mg per day in 3 divided doses
  Interventions: Drug: Gabapentin
- placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — gaba potentiating medication
  Other Names: neurontin
  Arms: Gabapentin
Drug: Placebo — a pill that looks exactly like the active medication but does not contain medication
  Other Names: Sugar Pill
  Arms: placebo

SUMMARY:
This treatment study is a 16-weeks outpatient clinical trial where subjects with alcohol dependence will get medication, which might help them to reduce or stop their drinking, or a placebo ( placebo is a capsule that looks the same as the investigational drug, but has no real medication. It is a "sugar pill").

DETAILED DESCRIPTION:
This treatment study is a 16-weeks outpatient clinical trial where subjects will get medication, which might help them to reduce or stop their drinking or a placebo ( placebo is a capsule that looks the same as the investigational drug, but has no real medication. It is a "sugar pill"). This study will recruit and randomize subjects who have expressed an interest in receiving treatment for alcohol dependence. Upon enrollment into this study there will be 11 outpatient visits. Each visit will last about 1-1.5 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Meets criteria for alcohol use disorder based on DSM-5 criteria
2. Meets criteria for history of alcohol withdrawal based on DSM-5 criteria
3. Able to maintain abstinence for a minimum of 3 days prior to randomization as verified by self report, urine ETG, and breathalyzer.

Exclusion Criteria:

1. Significant psychiatric or medical illness
2. No other substance abuse
3. Taking other medications known to treat alcohol use disorder
4. Unstable living arrangements
5. Significant legal problems pending

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-11; Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond F Anton, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Hoffman M, Voronin K, Book SW, Prisciandaro J, Bristol EJ, Anton RF. Sleep as an Important Target or Modifier in Alcohol Use Disorder Clinical Treatment: Example From a Recent Gabapentin Randomized Clinical Trial. J Addict Med. 2024 Sep-Oct 01;18(5):520-525. doi: 10.1097/ADM.0000000000001316. Epub 2024 May 31. PMID 38828963
- [Derived] Prisciandaro JJ, Hoffman M, Brown TR, Voronin K, Book S, Bristol E, Anton RF. Effects of Gabapentin on Dorsal Anterior Cingulate Cortex GABA and Glutamate Levels and Their Associations With Abstinence in Alcohol Use Disorder: A Randomized Clinical Trial. Am J Psychiatry. 2021 Sep 1;178(9):829-837. doi: 10.1176/appi.ajp.2021.20121757. Epub 2021 Jul 14. PMID 34256607
- [Derived] Anton RF, Latham P, Voronin K, Book S, Hoffman M, Prisciandaro J, Bristol E. Efficacy of Gabapentin for the Treatment of Alcohol Use Disorder in Patients With Alcohol Withdrawal Symptoms: A Randomized Clinical Trial. JAMA Intern Med. 2020 May 1;180(5):728-736. doi: 10.1001/jamainternmed.2020.0249. PMID 32150232

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The discrepancy of 6 participants is due to those subjects either violating protocol or not having evaluable data.
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 44 | 46
Completed | 31 | 28
Not Completed | 13 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 44 | 46 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (10.4) | 48.9 (9.9) | 49.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 34 | 35 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 41 | 44 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
% Heavy Drinking Days [Mean (Standard Deviation); unit: percent] — % heavy drinking days out of the 90 days reported via timeline followback. A heavy drinking day is defined as 4 or more drinks for females and 5 or more drinks for males in one day.
  percent | 82.9 (23) | 82.5 (21.6) | 82.7 (22.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With no Heavy Drinking Days (PSNHDD)
Description: The primary dependent variable will be the percent of subjects with no heavy drinking days (4 or more standard drinks for women and 5 or more standard drinks for men). Participants will report their daily alcohol use with using a daily calendar. No heavy drinking days is corrected for %dCDT.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 44 | 46
Participants | 12 | 4
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; This analysis compares between Gabapentin and Placebo, the number of individuals who reported no heavy drinking days throughout the entire trial, corrected for %dCDT; Test type: Superiority; p = .028, Regression, Logistic; This is the p-value output from the logistic regression model where medication group predicted the discrete variable for no heavy drinking days; Odds Ratio (OR) = 3.9

2. Secondary Outcome: Percent of Subjects With no Drinking Days (PSNDD)
Description: The secondary dependent variable will be percent of subjects with no drinking days (total abstinence). Participants will report their daily alcohol use with using a daily calendar. Abstinence is corrected for %dCDT.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 44 | 46
Participants | 8 | 2
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; This analysis compares between Gabapentin and Placebo, the number of individuals who reported no drinking days (abstinence) throughout the entire trial, corrected for %dCDT; Test type: Superiority; p = .053, Regression, Logistic; This is the p-value output from the logistic regression model where medication group predicted the discrete variable for abstinence; Odds Ratio (OR) = 4.9

3. Other Pre Specified Outcome: Number of Participants With No Drinking Days by AWS Score and Medication
Description: This analysis examines the interaction of medication group with a median split of the baseline Alcohol Withdrawal Scale (AWS) scores on the primary outcome variable (no heavy drinking days, corrected for %dCDT). Participants will report their daily alcohol use with using a daily calendar. AWS ranges from 0 to 44 where higher values correspond with more serious withdrawal (worse outcome).
Time Frame: 4 months
Population: The data for this analysis were split into two subgroups, based on the median split of AWS.
Measure: Count of Participants; unit: Participants
Groups:
- Low AWS/Gabapentin: Low on AWS median split variable, Gabapentin
- Low AWS/Placebo: Low on AWS median split variable, Placebo
- High AWS/Gabapentin: High on AWS median split variable, Gabapentin
- High AWS/Placebo: High on AWS median split variable, Placebo
Arm/Group | Low AWS/Gabapentin | Low AWS/Placebo | High AWS/Gabapentin | High AWS/Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
Participants | 2 | 3 | 10 | 1
Statistical Analysis 1: Comparison: High AWS/Gabapentin vs High AWS/Placebo; For the High AWS group, a chi squared analysis compares the number of individuals with no heavy drinking days between medication groups; Test type: Superiority; p = .001, Chi-squared
Statistical Analysis 2: Comparison: Low AWS/Gabapentin vs Low AWS/Placebo; For the Low AWS group, a chi squared analysis compares the number of individuals with no heavy drinking days between medication groups; Test type: Superiority; p = .67, Chi-squared

ADVERSE EVENTS:
Time Frame: Entire study - 16 weeks.
Description: Participants were evaluated via the SAFTEE interview 9 times throughout the 16 week period.
  We report the whole SAFTEE.
Arm/Group | Gabapentin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/46
Other Adverse Events (participants affected / at risk) | 44/44 | 44/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=44) | Placebo (N=46)
Abdominal Pain (Gastrointestinal disorders) | 10 (12) | 11 (16)
Decreased Appetite (General disorders) | 12 (18) | 11 (13)
Decreased Libido (General disorders) | 12 (24) | 5 (11)
Depression (Psychiatric disorders) | 24 (80) | 22 (60)
Diarrhea (Gastrointestinal disorders) | 23 (62) | 23 (42)
Dizziness (Nervous system disorders) | 25 (60) | 15 (27)
Fatigue (General disorders) | 30 (122) | 30 (108)
Headache (Nervous system disorders) | 32 (129) | 34 (89)
Increased Appetite (General disorders) | 23 (52) | 18 (32)
Increased Libido (General disorders) | 7 (8) | 4 (6)
Insomnia (General disorders) | 31 (92) | 33 (130)
Itching (Skin and subcutaneous tissue disorders) | 10 (26) | 9 (21)
Nausea (Gastrointestinal disorders) | 14 (26) | 18 (33)
Nervousness/Anxiety (Psychiatric disorders) | 35 (172) | 32 (127)
Rash (Skin and subcutaneous tissue disorders) | 7 (17) | 5 (7)
Somnolence (General disorders) | 6 (13) | 6 (7)
Suicidal Ideation (Psychiatric disorders) | 4 (12) | 2 (2)
Vomiting (Gastrointestinal disorders) | 9 (14) | 6 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT02349477/Prot_SAP_000.pdf